CLINICAL TRIAL: NCT00283855
Title: An Online Self Management Program for Adults With Rheumatoid Arthritis
Brief Title: RAHelp.Org: An Online Self Management Program for Adults With Rheumatoid Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Collaborators: U.S. Department of Education (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None
Other Study IDs: H133B031120-Proj 1
Record Dates: First submitted 2006-01-26; First posted 2006-01-30 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-09

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Self-Management; Internet
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (No Intervention): No intervention
- Online Self-Management (Active Comparator): RAHelp.org
  Interventions: Behavioral: Online Self-Management

INTERVENTIONS:
Behavioral: Online Self-Management — Online Self-Management
  Arms: Online Self-Management

SUMMARY:
The objective of this study is to determine the effects of an arthritis self-management program and an online support community delivered via an encrypted, secure web site on psychological well-being, pain, quality of life, global health status, and social supporting in adults with RA.

DETAILED DESCRIPTION:
Arthritis is the leading cause of disability in the United States. More than 7 million persons in this country report limitations in their daily activities due to arthritis. Rheumatoid arthritis alone affects 1 of every 100 persons in the US. Clinic-based self-management programs have been found to be effective in reducing both pain and disability for persons with RA. However, barriers to participation exist such as distance, time, limited transportation, and declining functional status. The Internet is widely used as a source of information about health issues and may provide an opportunity to reduce these barriers and extend consumer access to self-management approaches. It is necessary to determine the efficacy of Internet-delivered self-management programs.

ELIGIBILITY:
Inclusion Criteria:

* 18 or more years of age
* Rheumatoid Arthritis diagnosed by a rheumatologist
* Stable medication regimen for 3 months

Exclusion Criteria:

* Previous exposure to arthritis self-management programs
* Uncontrolled psychiatric comorbidity
* Uncontrolled medical comorbidity (e.g. active cancer)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2003-10; Primary Completion 2008-08 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Arthritis Impact Measurement Scales | baseline, 3 mos., 6 mos., 9 mos., 12 mos.

SECONDARY OUTCOMES:
Arthritis Self-Efficacy Scale | baseline, 3 mos., 6 mos., 9 mos., 12 mos
Rapid Assessment of Disease Activity in Rheumatology | baseline, 3 mos., 6 mos., 9 mos., 12 mos

OTHER OUTCOMES:
Social Provisions Scale | baseline, 3 mos., 6 mos., 9 mos., 12 mos
21-point Box Scale (a pain measure) | baseline, 3 mos., 6 mos., 9 mos., 12 mos
UCLA Loneliness Scale | baseline, 3 mos., 6 mos., 9 mos., 12 mos
Center for Epidemiological Studies - Depression Scale | baseline, 3 mos., 6 mos., 9 mos., 12 mos
Physical Activity Scale for the Elderly | baseline, 3 mos., 6 mos., 9 mos., 12 mos

CONTACTS AND LOCATIONS:
Overall Officials: Karen L Smarr, Ph.D., Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri-Columbia, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Smarr K; Musser D; Donovan Hanson K; Laffey J; Johnson R; Siva C; Parker J. Development of an online self-management intervention for persons with rheumatoid arthritis: The RAHelp.org project. Arthritis Rheum 2005 Sep;52(9):S718
- [Derived] Shigaki CL, Smarr KL, Siva C, Ge B, Musser D, Johnson R. RAHelp: an online intervention for individuals with rheumatoid arthritis. Arthritis Care Res (Hoboken). 2013 Oct;65(10):1573-81. doi: 10.1002/acr.22042. PMID 23666599